CLINICAL TRIAL: NCT02991300
Title: Open Label, Prospective, Consecutive Series Registry Database of BioPoly® RS Partial Resurfacing Patella Implant
Brief Title: BioPoly® RS Partial Resurfacing Patella Registry Study
Status: Completed | Type: Observational
Sponsor: BioPoly LLC (Industry)
Responsible Party: Sponsor
Other Study IDs: 1251001 V2.0
Record Dates: First submitted 2016-12-08; First posted 2016-12-13 (Estimated); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Cartilage Disease
Keywords: focal defect; focal lesion; chondral lesion; osteochondral lesion
MeSH Terms: conditions — Cartilage Diseases

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: BioPoly RS Partial Resurfacing Patella Implant

SUMMARY:
The data registry will increase the knowledge of outcomes for treatment of focal cartilage defects of the patella treated with the BioPoly RS Patella Implant and will allow monitoring of the clinical safety and performance of the device and surgical implantation kit

DETAILED DESCRIPTION:
The data registry will increase the knowledge of outcomes for treatment of focal cartilage defects of the patella treated with the BioPoly RS Patella Implant This study will also allow monitoring of the clinical safety and performance of the device and surgical implantation kit

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and older
* Cartilage lesion(s) located in the facets of the patella that have failed prior therapy (conservative or surgical)
* Symptomatic lesions classified as ICRS grade 2, 3, or 4
* Lesion size may not exceed 3.1 cm2 and must be circumscribed by a 15 mm or 20 mm circle of normal or nearly normal (ICRS Grade 0 or 1) cartilage, with an overall depth less than 4 mm from the articulating surface
* Subchondral bone quality sufficient to support the implant
* Understanding and willingness to comply with the post-operative rehabilitation instructions and follow-up visits.

Exclusion Criteria:

* Body mass index (BMI) ≥ 35
* Generalized degenerative or autoimmune arthritis
* Gout
* Uncorrected chronic malalignment of the patella (may be corrected at the same time as the implantation of the BioPoly device).
* Uncorrected ligamentous instability (may be corrected at the same time as the implantation of the BioPoly device).
* Kissing lesion on femur
* More than one implant required to accommodate lesion
* Allergy to ultra-high molecular weight polyethylene (UHMWPE), or hyaluronan/ hyaluronic acid (HA)
* Use with opposing articulating femoral components
* Any concomitant painful or disabling disease of the spine, hips, or lower limbs that would interfere with evaluation of the afflicted knee
* Pregnant, prisoner, vulnerable population, or unable to provide informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The population who will participate in this clinical study includes those patients 21 years of age or older who otherwise meet the inclusion/exclusion criteria.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2024-12 (Actual); Study Completion 2024-12 (Actual)

PRIMARY OUTCOMES:
KOOS Subscores | 2 year post-op
  KOOS
Kujala Anterior Knee Pain Scale | 2 year post-op
  Kujala
Medical Outcomes Study (SF-36) for generic "quality of life" | 2 years post-op
  SF-36
Activity using Tegner Score | 2 years post-op
  Tegner
Pain using VAS Pain | 2 years post-op
  VAS Pain

SECONDARY OUTCOMES:
Radiographic Assessment | Annually through 5 years post-op
  Radiographic Assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Nathwani, MD, Principal Investigator — Charing Cross Hospital
Locations (2):
- United Kingdom (2):
  - Charing Cross Hospital, London, England
  - Mid Yorkshire Hosp NHS, Wakefield

IPD SHARING:
Plan to Share IPD: No